CLINICAL TRIAL: NCT04669613
Title: Contrast Ultrasound Dispersion Imaging (CUDI) as a Diagnostic Modality in the Diagnosis of Renal Cell Carcinoma
Acronym: CUDI-RCC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, Prof.dr. H.P. Beerlage, Professor, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CUDI-RCC
Record Dates: First submitted 2020-07-21; First posted 2020-12-17 (Actual); Last update posted 2020-12-17 (Actual); Status verified 2020-12

CONDITIONS: Kidney Cancer
Keywords: Ultrasound; CEUS; CUDI; Contrast enhanced ultrasound; Contrast ultrasound dispersion imaging; Kidney cancer; renal cancer; carcinoma
MeSH Terms: conditions — Kidney Neoplasms; Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients (Experimental)
  Interventions: Other: CUDI

INTERVENTIONS:
Other: CUDI — Analysis of the CEUS data by means of Contrast ultrasound dispersion imaging
  Other Names: Contrast ultrasound dispersion imaging

SUMMARY:
Introduction The current limitations of renal cell carcinoma (RCC) imaging form a major deficit in the diagnostic pathway. Contrast Enhanced UltraSound (CEUS) has the potential to improve RCC detection and localization significantly. CEUS image interpretation is however difficult and subjective. To overcome these difficulties a CEUS quantification technique, Contrast-enhanced Ultrasound Dispersion Imaging (CUDI), has been developed in cooperation with the Eindhoven University of Technology (TU/e).

Study objective Primary objective: To assess the sensitivity and specificity of CUDI for recognizing malignant tissue in vivo.

Study population All patients scheduled for a partial or radial nephrectomy in the Amsterdam UMC (Amsterdam Universitair Medische Centra) Study Procedure This study is a prospective in-vivo study in patients scheduled for a partial or radical nephrectomy for a suspicious RCC in which we will perform CEUS imaging. The (partial) nephrectomy is part of standard care for patients with a suspicious lesion in the kidney. The additional ultrasound with infusion of an ultrasound contrast agent during ultrasound scanning is performed for the purpose of the study. CEUS imaging will be performed right before (partial) nephrectomy, with the patient being under general anesthesia. The CEUS and CUDI parametric maps will be interpreted by Investigator A in a blinded fashion with suspicious lesions each delineated. The (partial) nephrectomy will be performed by a qualified urologist, and the analysis of the histological specimens will be performed by a qualified pathologist. Sensitivity and specificity for CUDI will be calculated for all patients receiving a (partial) nephrectomy in which the tissue is sent for pathology.

Benefits Currently, most renal tumors are diagnosed by abdominal US, CT or MRI. Renal tumors are classified as cystic or solid lesions on imaging. The most important criteria for differentiating malignant lesions is the presence of enhancement after administration of contrast for CT or MRI in several different phases (4 phases CT-scan). Enhancement in renal masses is determined by comparing Hounsfield units before and after administration of contrast. A change of 15 or more Hounsfield units demonstrates enhancement. Specificity and sensitivity for detecting RCC are around 75% and 88% for CT, and around 89% and 87.5% for MRI, respectively.

Both CT and MRI can objectify a contrast-enhancing mass, suspicious for RCC, however, they cannot reliably distinguish a benign lesion (such as an oncocytoma or angiomyolipoma) from a malignant renal neoplasm. For that reason, patients are currently undergoing an RTB (renal tumor biopsy) to objectify pathology for deciding if treatment is necessary or not. Recent literature suggests up to 30% benign pathology after partial nephrectomy implicating overtreatment. RTB has been gradually introduced and increasingly used, however, an RTB is not without risks. Bleeding is the most documented complication. Recently even tumor tract seeding has been under discussion. Improving imaging by using CUDI for differentiating benign from malignant lesions instead of performing an RTB could prevent those risks for patients.

Risk assessment There is a small risk of contrast-related adverse events (AE) for participants. After use in millions of patients, AE to the ultrasound contrast agent appear to be transient, mild and rare, and mostly consist of transient alteration of taste, local pain at the injection site and facial or general flush. In some cases, a mild allergic reaction is described. Patients will be informed of the risk during contrast exposure, and it will be described in the patient information file.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18 years
* signed informed consent
* scheduled for a radical- or partial nephrectomy for the suspicious of a renal tumor.

Exclusion Criteria:

* Earlier treatment of renal masses
* History of any clinically evidence of cardiac right-to-left shunts
* Severe pulmonary hypertension (pulmonary artery pressure >90 mmHg) or uncontrolled systemic hypertension or respiratory distress syndrome
* Has any medical condition or other circumstances which would significantly decrease the chances of obtaining reliable data, achieving study objectives, or completing the study
* Is incapable of understanding the language in which the information for the patient is given
* Tumor cannot be visualized/localized on ultrasound imaging
* Previous hypersensitivity allergic reactions
* Known allergy of macrogol 4000, distearoylphosphatidylcholine, dipalmitoylphosphatidylglycerol Sodium, Palmitic acid
* Use of dobutamine or conditions suggesting cardiovascular instability where dobutamine is contraindicated.
* Pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2020-12-30 (Estimated); Primary Completion 2021-01-01 (Estimated); Study Completion 2021-04-01 (Estimated)

PRIMARY OUTCOMES:
per-patient RCC detection rates | through study completion, an average of 1 year
Rate of malignant histology that can be correlated to CUDI-parameters | through study completion, an average of 1 year
  After receiving both the CUDI-data and the histology data, both will be compared to check if the regions that show different CUDI-parameters match the regions with malignancy in histology
Wash out time as a parameter to measure the dispersion of the micro bubbles of the CUDI contrast agent | through study completion, an average of 1 year
  This is a physical parameter that is quantified from CEUS-data by CUDI. The wash out time is the time that it takes for the micro bubbles to disappear.

SECONDARY OUTCOMES:
sensitivity of CUDI | through study completion, an average of 1 year
specificity of CUDI | through study completion, an average of 1 year
negative predictive value of CUDI | through study completion, an average of 1 year
positive predictive value of CUDI | through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Amsterdam UMC, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ljungberg B, Bensalah K, Canfield S, Dabestani S, Hofmann F, Hora M, Kuczyk MA, Lam T, Marconi L, Merseburger AS, Mulders P, Powles T, Staehler M, Volpe A, Bex A. EAU guidelines on renal cell carcinoma: 2014 update. Eur Urol. 2015 May;67(5):913-24. doi: 10.1016/j.eururo.2015.01.005. Epub 2015 Jan 21. PMID 25616710
- [Result] Israel GM, Bosniak MA. Pitfalls in renal mass evaluation and how to avoid them. Radiographics. 2008 Sep-Oct;28(5):1325-38. doi: 10.1148/rg.285075744. PMID 18794310
- [Result] Vogel C, Ziegelmuller B, Ljungberg B, Bensalah K, Bex A, Canfield S, Giles RH, Hora M, Kuczyk MA, Merseburger AS, Powles T, Albiges L, Stewart F, Volpe A, Graser A, Schlemmer M, Yuan C, Lam T, Staehler M. Imaging in Suspected Renal-Cell Carcinoma: Systematic Review. Clin Genitourin Cancer. 2019 Apr;17(2):e345-e355. doi: 10.1016/j.clgc.2018.07.024. Epub 2018 Aug 11. PMID 30528378
- [Result] Fernando A, Fowler S, O'Brien T; British Association of Urological Surgeons (BAUS). Nephron-sparing surgery across a nation - outcomes from the British Association of Urological Surgeons 2012 national partial nephrectomy audit. BJU Int. 2016 Jun;117(6):874-82. doi: 10.1111/bju.13353. Epub 2015 Nov 18. PMID 26469291
- [Result] Marconi L, Dabestani S, Lam TB, Hofmann F, Stewart F, Norrie J, Bex A, Bensalah K, Canfield SE, Hora M, Kuczyk MA, Merseburger AS, Mulders PFA, Powles T, Staehler M, Ljungberg B, Volpe A. Systematic Review and Meta-analysis of Diagnostic Accuracy of Percutaneous Renal Tumour Biopsy. Eur Urol. 2016 Apr;69(4):660-673. doi: 10.1016/j.eururo.2015.07.072. Epub 2015 Aug 29. PMID 26323946
- [Result] Macklin PS, Sullivan ME, Tapping CR, Cranston DW, Webster GM, Roberts ISD, Verrill CL, Browning L. Tumour Seeding in the Tract of Percutaneous Renal Tumour Biopsy: A Report on Seven Cases from a UK Tertiary Referral Centre. Eur Urol. 2019 May;75(5):861-867. doi: 10.1016/j.eururo.2018.12.011. Epub 2018 Dec 24. PMID 30591353